CLINICAL TRIAL: NCT03405389
Title: An International, Multicenter, Focused Registry to Collect Clinical Data on the MatrixWAVE Mandibulo-Maxillary Fixation System
Brief Title: Focused Registry to Collect Clinical Data on the MatrixWAVE System
Acronym: MatrixWAVE
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: FR_MatrixWave
Record Dates: First submitted 2018-01-11; First posted 2018-01-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mandibular Fractures
Keywords: mandibulo-maxillary fixation; malocclusion
MeSH Terms: conditions — Mandibular Fractures; Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients diagnosis of a mandibular fracture requiring Open Reduction and Internal Fixation (ORIF) and use of Mandibulo-Maxillary fixation (MMF) during or subsequent to surgical intervention for a minimum of two weeks
  Interventions: Procedure: MatrixWAVE MMF System

INTERVENTIONS:
Procedure: MatrixWAVE MMF System — Standard of care treatment of the injury and use of the MatrixWAVE MMF system to establish occlusion

SUMMARY:
The goal of this registry is to evaluate the performance of the MatrixWAVE(TM) MMF system in patients suffering from non-condylar and/or condylar fractures. The evaluation will focus on the clinical performance in terms of :

* surgical technique
* application time
* intra- and postoperative complications
* short term patient-reported outcomes

DETAILED DESCRIPTION:
Following standard of care (routine) procedures, a total number of 50 patients suffering from non-condylar and/or condylar fractures of the mandible requiring MMF for a minimum of two weeks during or subsequent to open reduction internal fixation (ORIF) will be prospectively enrolled in this registry.

Data on the classification of the injury (AO CMF fracture classification system) and the time needed for application of the MatrixWAVE(TM) MMF system will be collected.

Follow-up (FU) visits will be performed between 2 to 6 weeks and at 3 months according to standard of care to evaluate the mandible function impairment, pain and local complications (anticipated procedure-related adverse events) related to the MatrixWAVE(TM) MMF system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of the surgery
* Diagnosis of a mandibular fracture requiring ORIF and use of MMF during or subsequent to surgical intervention for a minimum of two weeks
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the clinical investigation according to the Registry Plan (RP)
  * Signed and dated EC/IRB approved written informed consent

Exclusion Criteria:

* Pre-traumatic non-occlusion due to hypodontia, edentulousness or severe malalignment of dental arches (e.g. complete crossbite)
* Concomitant maxillary fracture (e.g. Le Fort)
* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the registry period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present registry
* Intra-operative decision of the surgeon to use other MMF systems than the MatrixWAVE MMF system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old suffering with a mandibilar fracture without involvement of the condyle(s) or maxilla.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Time of application | Intraoperative
  Time required by the surgeons to apply the MatrixWAVE MMF system

SECONDARY OUTCOMES:
Patient-reported outcome (Likert scale) | 6 weeks
  Effect of MatrixWAVE MMF system on daily-life activities (speaking, eating and chewing, kissing)

CONTACTS AND LOCATIONS:
Overall Officials: Paris Liokatis, Dr. med., Principal Investigator — Klinikum der Universität München
Locations (2):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Ludwig-Maximillians University, München, Germany

IPD SHARING:
Plan to Share IPD: No